CLINICAL TRIAL: NCT00651924
Title: Piloting Interactive Voice Response Modules for Chronic Pain Treatment
Brief Title: Piloting IVR (Interactive Voice Response) for Chronic Pain Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SHP 08-147
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Pain
Keywords: chronic pain; IVR; cognitive-behavior therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (No Intervention): Review the materials and provide feedback regarding how understandable, engaging, and informative the materials are
- Phase 2 (Experimental): Piloting the 'IVR-based Cognitive-behavior therapy' using the new materials
  Interventions: Behavioral: IVR-based Cognitive-behavior therapy

INTERVENTIONS:
Behavioral: IVR-based Cognitive-behavior therapy — Standard cognitive-behavior therapy for chronic pain management using Interactive Voice Response (IVR) compatible materials and handouts
  Arms: Phase 2

SUMMARY:
This study is designed to develop and test the use of Interactive Voice Response (IVR) technology to deliver pain management treatment. IVR allows individuals to receive and provide information by using their touchtone telephone. This will allow more people with chronic pain to receive treatment even if they are not able to drive to an appointment regularly. In the first part of the study, the investigators will develop new materials like patient handbooks and pre-recorded explanations about common pain control techniques. In the second part of the study, a small number of persons with chronic pain will receive treatment using the new materials. We will ask for their feedback about how well they liked using the new materials and if the materials are understandable. This will allow us to revise the materials if we need to prior to studying them with a larger group of people with chronic pain.

DETAILED DESCRIPTION:
Background:

Cognitive behavioral therapy (CBT) has been shown in two meta-analyses to be effective in reducing pain intensity, disability, and affective distress in persons with chronic pain. Although effective, traditional CBT is time-intensive and requires patients to make frequent office visits. An alternative is to improve treatment accessibility and efficiency of treatment provision through the use of electronic methods such as interactive voice response (IVR) technology.

Objectives:

This pilot project was designed to test the feasibility and perceived value of IVR-based CBT intervention materials for the treatment of chronic pain. The project involved adapting traditional CBT materials for use in a IVR-based chronic pain treatment.

Methods:

The project occurred in two phases. Phase 1 included the revision of materials to support the IVR-based intervention including 1) a patient handbook, 2) a library of IVR-compatible scripts for the presentation of pain treatment topics, and 3) guidelines for providing personalized feedback. Phase 2 included the evaluation of the developed materials by a small group of patients with chronic pain. After the treatment materials were revised, their usability, feasibility and perceived value were tested with a small sample of Veterans with chronic pain.

Status:

This study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Pain for at least 6 months;
* Average pain level of >3 on a scale of 0 (no pain) to 10 (worst imaginable);
* Access to touchtone phone

Exclusion Criteria:

* Current alcohol or substance abuse;
* Current psychosis;
* Current suicidal ideation;
* Current life threatening or acute physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Kerns, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited Dec. 2008-May 2012 for all phases. Participants were recruited from a Comprehensive Pain Clinic and through provider referral.
Groups:
- Phase 1: Review of materials and provide feedback regarding how understandable, engaging, and informative the materials are. Revisions will be made based on this feedback.
- Phase 2: Undergo IVR-based Cognitive Behavioral Therapy treatment using the new materials.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 18 | 9
Completed | 18 | 2
Not Completed | 0 | 7
Not completed — Withdrawal by PI | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: Phase 2: two individuals completed all 10 sessions of treatment, however, we have baseline measures on 6 individuals (1 dropped after 5 sessions, 2 dropped after 1 session, 1 dropped after 2 sessions and 1 dropped after 4 sessions).
Groups:
- Phase 2: Pilot IVR-based Cognitive-behavior therapy: Standard cognitive-behavior therapy for chronic pain management using Interactive Voice Response (IVR) compatible materials and handouts
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8.25) | 56 (17) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 17 | 6 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11 | 6 | 17
  Black | 6 | 0 | 6
  Hispanic | 1 | 0 | 1
Pain Severity [Mean (Standard Deviation); unit: units on a scale] — 10 point likert scale: 0 No Pain at All - 10 Worst Pain Imaginable
  Missing data for 11 patients (Phase 1- 9; Phase 2 - 2)
  units on a scale | 6.33 (1.77) | 5.88 (0.63) | 6.21 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Comprehension
Description: Each treatment session had 5 True / False questions that corresponded with the material in the patient handbook. Phase 1 participants reviewed individual treatment modules in the patient handbook to provide immediate feedback regarding how understandable, engaging, and informative they find the materials. Phase 2 participants' used the patient materials as part of treatment and the true/false questions were used to evaluate comprehension of the materials. Example questions: Chronic pain can affect how you feel physically and emotionally (T); Relaxation is the same as being lazy and unproductive (F).
Time Frame: Immediately after review of materials (phase 1); 1 week post review of materials (phase 2)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Percent of questions answered correctly
Groups:
- Phase 1: Qualitative interviews
- Phase 2: Pilot IVR-based CBT treatment
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 18 | 5
Percent of questions answered correctly | 92.14 (12.51) | 96.42 (9.29)

ADVERSE EVENTS:
Time Frame: 12/02/2008 - 01/21/2011]
Groups:
- Phase 1: Review of newly created materials and provide feedback regarding how understandable, engaging, and informative the materials are.
- Phase 2: Pilot the newly developed materials during a 10-week course of cognitive behavioral therapy for chronic pain
Arm/Group | Phase 1 | Phase 2
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 0/18 | 0/9

LIMITATIONS AND CAVEATS:
Difficulty recruiting for phase 2 lead to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No